CLINICAL TRIAL: NCT04219618
Title: The Left Ventricular Assist Device Off or On Pump Implantation Study: A Single-center Randomized Trial (LVAD-ON-OFF)
Brief Title: The Left Ventricular Assist Device (LVAD) Off or On Pump Implantation Study
Acronym: LVAD-ON-OFF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because the manufacturer stopped producing the HeartWare LVAD device.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Igor Gregoric, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0926
Record Dates: First submitted 2019-12-11; First posted 2020-01-07 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; LVAD
Keywords: LVAD
MeSH Terms: conditions — Heart Failure | interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Off-Pump (Experimental)
  Interventions: Device: Off-Pump
- On-Pump (Active Comparator)
  Interventions: Device: On-Pump

INTERVENTIONS:
Device: Off-Pump — After a standard median sternotomy, pericardium will be divided to expose the heart and major vessels, and the aortic cannulation sutures will be placed. Pyramid positioner will be applied to the apex of the heart, and the heart will be manually elevated upward. The inflow cannula placement location and placement of the sewing ring will be done with pledged sutures. The LV diaphragmatic site coring will be completed, and immediate LV digital exploration will be accomplished. The LVAD inflow cannula will be inserted through the sewing ring into the LV cavity. Upon completing proper LVAD inflow cannula placement into the LV and securing it in position, the heart will be dropped into the pericardial cavity with the outflow graft elevated for LVAD and outflow graft de-airing and to prevent potential later air embolization. A partial occlusion clamp will be placed on the ascending aorta and appropriately trimmed outflow graft will be sewn to the aorta.
  Arms: Off-Pump
Device: On-Pump — A standard median sternotomy incision will be performed and pericardium divided to expose the heart and major vessels. Cannulation will be done through the aorta and the right atrium and the patient will be put on cardiopulmonary bypass (CPB). The patient's heart will be freed from the surrounding tissues. With a cylindrical blade, the surgeon will excise a core of myocardium from the apex. The LVAD sewing ring will then be sutured to the margins of the apical hole. The LVAD will be inserted into the LV cavity through the sewing ring. The outflow graft will be measured for the anastomosis into the aortic root. Partial occlusion clamp will be placed on the aortic root and the anastomosis will be performed. De-airing will be performed and the LVAD will be started. The patient will then be weaned from CPB and decannulated.
  Arms: On-Pump

SUMMARY:
The purpose of this study is to compare adverse events after off-pump LVAD surgery or on-pump LVAD surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient has had a diagnosis of end stage heart failure, New York Heart association (NYHA) class III or IV HF for a minimum of 90 days prior to screening.
* The patient has guideline-directed medical therapy according to American College of Cardiology(ACC)/American Heart Association (AHA)/European Society of Cardiology(ESC) heart failure(HF) guidelines
* The patient has an Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) score of 1-3.
* Left ventricular assist device (LVAD) placement is intended as a bridge to transplant (BTT) or destination therapy (DT) with either HeartWare Ventricular Assist Device (HVAD) or HeartMate III LVAD.
* The patient is able to sign informed consent form and Release of Medical Information Form.
* The patients is willing and able to participate in scheduled follow-up appointments.

Exclusion Criteria:

* The patient requires concomitant surgery for left ventricular or atrial appendage closure or the patient has severe aortic insufficiency, mitral stenosis, or severe tricuspid regurgitation.
* The patient has an intracardiac thrombus or other mass diagnosed by echocardiography, left ventriculogram, or other imaging.
* Planned insertion of right ventricular(RV) support device (either temporary or permanent).
* The patient has suffered an acute cardiovascular event such as acute coronary syndrome (ST elevation myocardial infarction (STEMI) or Non-ST elevation myocardial infarction (NSTEMI), or unstable angina, or underwent any cardiac surgery or interventional cardiac or peripheral vascular procedure within 30 days prior to LVAD implantation.
* The patient has had ischemic or hemorrhagic stroke as diagnosed by CT or MRI within 90 days prior to study enrollment.
* The patient had prior heart or other organ transplantation, or surgically implanted LVAD or cardiac shunt.
* The patient will likely need an immediate heart transplant due to hemodynamic instability.
* The patient has had a known active malignancy or treatment for cancer within the past year except for localized prostate cancer, cervical carcinoma in situ, breast cancer in situ, or non-melanoma skin cancer that has been definitively treated.
* The patient has history of any malignancy where expected survival is less than two years. Past medical history of cancer is not exclusionary as long as subject has been disease-free for at least one years since the time of diagnosis and treatment.
* Patient has a severe co-morbidity (current need for hemodialysis or current glomerular filtration rate(GFR) ≤20 mL/minute/1.73 m2 estimated by Modification of Diet in Renal Disease( MDRD)calculation; hepatic impairment defined as liver function tests [alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)] >3x Upper Limit of Normal within 30 days prior to LVAD implantation or known objectively confirmed intrinsic liver disease (e.g., cirrhosis, chronic hepatitis B or hepatitis C virus infection)).
* The patient has a known bleeding diathesis or thrombocytopenia defined as platelet count <50,000 platelets/μL.
* The patient has peri/postpartum cardiomyopathy, or is a pregnant or lactating woman, or a woman of child-bearing age not using a suitable method of contraception.
* The patient, who in the absence of an Implantable Cardioverter Defibrillator (ICD) (or any implanted device capable of defibrillation), has a history of malignant ventricular arrhythmia or sustained ventricular tachycardia (VT), with sustained VT demonstrated by Q wave R wave S wave (QRS) complexes wider than 120 milliseconds, lasting more than 30 seconds, and with a rate of more than 100 beats per minute on screening ECG or other data supporting this diagnosis.
* Recent history of psychiatric disease, including drug or alcohol abuse, that is likely to impair, in the opinion of the investigator, the subject's ability to comply with protocol-mandated procedures.
* Participation in any other clinical investigation that is likely to confound study results or affect study outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor D Gregoric, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On-Pump | Off-Pump
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Pump | Off-Pump | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (0) | 39 (0) | 39 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Composite Outcome of Moderate or Severe Right Ventricular (RV) Dysfunction (Perioperative Right Heart Failure), Severe Renal Dysfunction Requiring Renal Replacement Therapy, Thrombotic Complications, or Death From Any Cause
Description: Perioperative right ventricular (RV) failure is defined by the Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) scoring as the need for intravenous inotropes for >14 days post-operatively or a right ventricular assist device (RVAD). RV function will be measured by tricuspid annular plane systolic excursion (TAPSE) values assessed using echocardiography. Additionally, hemodynamic evidence of RV dysfunction will also be collected with: a right-atrial pressure (RAP): pulmonary capillary wedge pressure (PCWP) ratio of ≥ 0.67.
  A thrombotic complication is defined as any thromboembolic event (transient ischemic attack or stroke objectively confirmed with computed tomography) or confirmed pump thrombus.
Time Frame: from time of implantation to 30 days post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With a Need for Blood Product Transfusion Within 48-hours Post-implantation
Time Frame: from time of implantation to 48 hours post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

3. Secondary Outcome: Operative Safety as Indicated by the Number of Participants Who Died Within 30 Days Post-implantation
Time Frame: from time of implantation to 30 days post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Operative Safety as Indicated by Chest Tube Output Within 24 Hours of Implantation
Time Frame: from time of implantation to 24 hours post-implantation
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
milliliters (mL) | 180 (0) | 100 (0)

5. Secondary Outcome: Operative Safety as Indicated by Number of Participants Who Underwent Post-operative Re-exploration for Bleeding
Time Frame: from time of implantation to 30 days post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Allosensitization
Description: Allosensitization is defined as calculated panel reactive antibody (cPRA) greater than 10%.
Time Frame: 30 days post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Allosensitization
Description: Allosensitization is defined as calculated panel reactive antibody (cPRA) greater than 10%.
Time Frame: 6 months post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Allosensitization
Description: Allosensitization is defined as calculated panel reactive antibody (cPRA) greater than 10%.
Time Frame: 12 months post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Readmissions for Heart Failure
Time Frame: from time of implantation to 1 year post-implantation
Measure: Number; unit: readmissions
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
readmissions | 2 | 0

10. Secondary Outcome: Overall Hemostatic Potential
Time Frame: Baseline
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Overall Coagulation Potential
Time Frame: Baseline
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Overall Fibrinolytic Potential
Time Frame: Baseline
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Overall Hemostatic Potential
Time Frame: 48 hours post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Overall Coagulation Potential
Time Frame: 48 hours post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Overall Fibrinolytic Potential
Time Frame: 48 hours post-implantation
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With Major Bleeding
Description: Major bleeding is defined as an episode of suspected internal or external bleeding that results in one or more of the following: death, re-operation, hospitalization, transfusion of red blood cells according to INTERMACS definition.
Time Frame: 30 days post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Major Bleeding
Description: as for outcome 16
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Major Bleeding
Description: as for outcome 16
Time Frame: 12 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Off-Pump | On-Pump
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Early termination was necessary because the manufacturer stopped producing the LVAD device, so the study wasn't feasible anymore.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04219618/Prot_SAP_000.pdf